CLINICAL TRIAL: NCT00875277
Title: A Psoriasis Plaque Test Comparing LEO 29102 Cream and Its Different Combinations to Daivobet® Ointment and a Vehicle Control for the Treatment of Psoriasis Vulgaris
Brief Title: A Psoriasis Plaque Test With LEO 29102 Cream and Its Combination Products
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PLQ-003
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — 2-(6-(2-(3,5-dichloro-4-pyridyl)acetyl)-2,3-dimethoxyphenoxy)-N-propylacetamide; betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LEO 29102 cream (Experimental): LEO 29102 2.5 mg/g cream applied topically twice daily for 4 weeks
  Interventions: Drug: LEO 29102 cream
- LEO 29102 Cream Vehicle (Placebo Comparator): LEO 29102 cream vehicle applied topically twice daily for 4 weeks.
  Interventions: Drug: LEO 29102 Cream Vehicle
- Betamethasone Dipropionate Cream (Experimental): Betamethasone 0.5 mg/g (as dipropionate) cream applied topically twice daily for 4 weeks.
  Interventions: Drug: Betamethasone Dipropionate Cream
- LEO 29102 Plus Calcipotriol Cream (Experimental): LEO 29102 2.5 mg/g plus calcipotriol 50mcg/g cream applied topically twice daily for 4 weeks.
  Interventions: Drug: LEO 29102 Plus Calcipotriol Cream
- LEO 29102 Plus Betamethasone Dipropionate (Experimental): LEO 29102 2.5 mg/g plus betamethasone 0.5 mg/g (as dipropionate) cream applied topically twice daily for 4 weeks.
  Interventions: Drug: LEO 29102 Plus Betamethasone Dipropionate
- Daivobet® Ointment (Active Comparator): Daivobet® ointment, combination of calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) applied topically twice daily for 4 weeks.
  Interventions: Drug: Daivobet® Ointment

INTERVENTIONS:
Drug: LEO 29102 cream
  Arms: LEO 29102 cream
Drug: LEO 29102 Cream Vehicle
  Arms: LEO 29102 Cream Vehicle
Drug: Betamethasone Dipropionate Cream
  Arms: Betamethasone Dipropionate Cream
Drug: LEO 29102 Plus Calcipotriol Cream
  Arms: LEO 29102 Plus Calcipotriol Cream
Drug: LEO 29102 Plus Betamethasone Dipropionate
  Arms: LEO 29102 Plus Betamethasone Dipropionate
Drug: Daivobet® Ointment
  Arms: Daivobet® Ointment

SUMMARY:
The purpose of this trial is to evaluate the anti-psoriatic effect of LEO 29102 cream and its combination with calcipotriol and betamethasone using a psoriasis plaque test method.

ELIGIBILITY:
Inclusion Criteria: (in summary)

* Subjects having understood and signed an informed consent form
* All skin types
* Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs or trunk. The lesions must have a total size suitable for application. The subjects should be asked if their lesions have been stable
* Subjects willing and able to follow all the study procedures and complete the whole study
* Subjects affiliated to social security system

Exclusion Criteria: (in summary)

* Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding
* Subjects using biological therapies (marketed or not marketed) with a possible effect on psoriasis (e.g. alefacept, efalizumab, etanercept, infliximab, adalimumab) within 12 weeks prior to study drug administration
* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D-analogues, retinoids, immunosuppressants) within the 4-week period prior to randomisation
* Subjects using one of the following topical drugs for the treatment of psoriasis within four (4) weeks prior to study drug administration: - Potent or very potent (WHO group III-IV) corticosteroids - PUVA or Grenz ray therapy
* Subjects using one of the following topical drugs for the treatment of psoriasis within two (2) weeks prior to study drug administration: - WHO group I-II corticosteroids - Topical retinoids - Vitamin D-analogues - Topical immunomodulators (e.g. macrolides) - Anthracen derivatives - Tar - Salicylic acid - UVB therapy
* Subjects with skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds within the plaque test areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, International Clinical Development, MD, Study Director — LEO Pharma
Locations (1):
- LEO Pharma site, Saint-Quentin-en-Yvelines, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were treated with the investigational medicinal products for 4 weeks followed by a 10-day follow-up period.
Groups:
- All Randomized Participants: All randomized participants received the six investigational medicinal products on six different test sites. LEO 29102 cream, LEO 29102 plus calcipotriol cream, LEO 29102 plus betamethasone dipropionate cream, Daivobet® ointment, Betamethasone dipropionate cream, and LEO 29102 cream vehicle applied topically once daily six times a week for 4 weeks (not on Sundays) on six different 2-cm diameter site (one per study preparation).
Period: Overall Study
Arm/Group | All Randomized Participants
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants received the six products on six different test sites.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Region of Enrollment [Number; unit: participants]
  France | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Clinical Score (TCS) of the Clinical Symptoms Compared to Baseline (Day 1)
Description: The (sub)investigator made the following clinical assessments by use of the scale below:
  Score; Intensity; Description
  Erythema:
  0; No evidence; Normal skin color 0.5; Doubtful or very mild 1.0; Mild; Pink light red 1.5; Mild to moderate 2.0; Moderate; Red 2.5; Moderate to severe 3.0; Severe; Intense red
  Scaling:
  0; No evidence; No scaling 0.5; Doubtful or very mild 1.0; Mild; Slight roughness, mainly fine scales 1.5; Mild to moderate 2.0; Moderate; Coarse scaling 2.5; Moderate to severe 3.0; Severe; Coarse, thick scales
  Infiltration:
  0; No evidence 0.5; Doubtful or very mild 1.0; Mild Slight definite infiltration 1.5; Mild to moderate 2.0; Moderate; Moderate infiltration 2.5; Moderate to severe 3.0; Severe; Very marked infiltration
  The TCS was defined as the sum of erythema plus scaling plus thickness scores. The TCS therefore ranged from 0 (all symptoms absent) to 9 (all symptoms severe).
Time Frame: From baseline (Day 1) to end of treatment (Day 29)
Population: The 24 participants that were randomized received all products distributed on six different test sites on the body.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale | -1.60 (1.18) | -4.96 (1.99) | -3.04 (1.34) | -3.96 (1.49) | -5.56 (1.28) | -6.10 (1.06)
Statistical Analysis 1: Comparison: LEO 29102 Cream Vehicle vs Betamethasone Dipropionate Cream; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: LEO 29102 Cream Vehicle vs LEO 29102 Cream; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: LEO 29102 Cream Vehicle vs LEO 29102 Plus Calcipotriol Cream; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: LEO 29102 Cream Vehicle vs LEO 29102 Plus Betamethasone Dipropionate; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: LEO 29102 Cream Vehicle vs Daivobet® Ointment; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 6: Comparison: Betamethasone Dipropionate Cream vs LEO 29102 Cream; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 7: Comparison: Betamethasone Dipropionate Cream vs LEO 29102 Plus Calcipotriol Cream; Test type: Superiority; p = 0.035, t-test, 2 sided
Statistical Analysis 8: Comparison: Betamethasone Dipropionate Cream vs LEO 29102 Plus Betamethasone Dipropionate; Test type: Superiority; p = 0.082, t-test, 2 sided
Statistical Analysis 9: Comparison: Betamethasone Dipropionate Cream vs Daivobet® Ointment; Test type: Superiority; p = 0.009, t-test, 2 sided
Statistical Analysis 10: Comparison: LEO 29102 Cream vs LEO 29102 Plus Calcipotriol Cream; Test type: Superiority; p = 0.012, t-test, 2 sided
Statistical Analysis 11: Comparison: LEO 29102 Cream vs LEO 29102 Plus Betamethasone Dipropionate; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 12: Comparison: LEO 29102 Cream vs Daivobet® Ointment; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 13: Comparison: LEO 29102 Plus Calcipotriol Cream vs LEO 29102 Plus Betamethasone Dipropionate; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 14: Comparison: LEO 29102 Plus Calcipotriol Cream vs Daivobet® Ointment; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 15: Comparison: LEO 29102 Plus Betamethasone Dipropionate vs Daivobet® Ointment; Test type: Superiority; p = 0.089, t-test, 2 sided

2. Secondary Outcome: Change in Single Clinical Symptom Score: Erythema, Scaling, Infiltration Compared to Baseline
Description: as for outcome 1
Time Frame: From baseline (Day 1) to end of treatment (Day 29)
Population: The 24 participants that were randomized received all products distributed on six different test sites on the body.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale
  Erythema | -0.42 (0.48) | -1.71 (0.81) | -0.90 (0.55) | -1.19 (0.70) | -1.85 (0.63) | -1.88 (0.45)
  Infiltration | -0.46 (0.33) | -1.46 (0.75) | -0.85 (0.52) | -1.17 (0.50) | -1.75 (0.53) | -2.04 (0.55)
  Scaliness | -0.73 (0.57) | -1.79 (0.62) | -1.29 (0.51) | -1.60 (0.55) | -1.96 (0.41) | -2.19 (0.41)

3. Secondary Outcome: Change in Erythema Compared to Baseline
Description: The severity of the symptoms was rated on screening and on study Days 1 (baseline), 4, 8, 11, 15, 18, 22, 25 and 29 (end of treatment) according to the 0-3 with half-point TCS grading scale.
  The (sub)investigator made the following clinical assessments by use of the scale below:
  Score; Intensity; Description
  Erythema:
  0; No evidence; Normal skin color 0.5; Doubtful or very mild 1.0; Mild; Pink light red 1.5; Mild to moderate 2.0; Moderate; Red 2.5; Moderate to severe 3.0; Severe; Intense red
Time Frame: At Day 4, Day 8, Day 11, Day 15, Day 18, Day 22 and Day 25
Population: The 24 participants that were randomized received all products distributed on six different test sites on the body.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  Visit 5 (Day 4) | -0.04 (0.25) | -0.21 (0.29) | -0.02 (0.18) | -0.08 (0.24) | -0.40 (0.42) | -0.38 (0.42)
  Visit 8 (Day 8) | -0.08 (0.38) | -0.67 (0.46) | -0.31 (0.32) | -0.29 (0.29) | -0.92 (0.43) | -0.88 (0.56)
  Visit 11 (Day 11) | -0.23 (0.33) | -0.94 (0.47) | -0.46 (0.33) | -0.44 (0.37) | -1.17 (0.43) | -1.19 (0.66)
  Visit 14 (Day 15) | -0.40 (0.36) | -1.23 (0.69) | -0.60 (0.36) | -0.77 (0.42) | -1.46 (0.59) | -1.40 (0.66)
  Visit 17 (Day 18) | -0.44 (0.40) | -1.33 (0.76) | -0.75 (0.42) | -0.98 (0.40) | -1.71 (0.61) | -1.63 (0.56)
  Visit 20 (Day 22) | -0.46 (0.49) | -1.48 (0.80) | -0.83 (0.55) | -1.04 (0.51) | -1.75 (0.66) | -1.85 (0.60)
  Visit 23 (Day 25) | -0.42 (0.43) | -1.54 (0.81) | -0.85 (0.54) | -1.08 (0.50) | -1.83 (0.72) | -1.94 (0.54)

4. Secondary Outcome: Change in Scaling Compared to Baseline
Description: The severity of the symptoms was rated on screening and on study Days 1 (baseline), 4, 8, 11, 15, 18, 22, 25 and 29 (end of treatment) according to the 0-3 with half-point TCS grading scale.
  The (sub)investigator made the following clinical assessments by use of the scale below:
  Score; Intensity; Description
  Scaling:
  0; No evidence; No scaling 0.5; Doubtful or very mild 1.0; Mild; Slight roughness, mainly fine scales 1.5; Mild to moderate 2.0; Moderate; Coarse scaling 2.5; Moderate to severe 3.0; Severe; Coarse, thick scales
Time Frame: At Day 4, Day 8, Day 11, Day 15, Day 18, Day 22, and Day 25
Population: The 24 participants that were randomized received all products distributed on six different test sites on the body.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LEO 29102 Plus Calcipotriol Cream: LEO 29102 2.5 mg/g plus calcipotriol 50 mcg/g cream applied topically twice daily for 4 weeks.
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  Visit 5 (Day 4) | -0.17 (0.35) | -0.31 (0.41) | -0.13 (0.30) | -0.21 (0.41) | -0.33 (0.43) | -0.52 (0.38)
  Visit 8 (Day 8) | -0.27 (0.42) | -0.88 (0.61) | -0.44 (0.58) | -0.63 (0.58) | -1.17 (0.67) | -1.19 (0.48)
  Visit 11 (Day 11) | -0.40 (0.33) | -1.15 (0.54) | -0.63 (0.42) | -0.71 (0.61) | -1.48 (0.58) | -1.92 (0.55)
  Visit 14 (Day 15) | -0.52 (0.52) | -1.33 (0.64) | -0.73 (0.47) | -1.00 (0.55) | -1.67 (0.58) | -2.04 (0.49)
  Visit 17 (Day 18) | -0.65 (0.45) | -1.56 (0.60) | -0.90 (0.47) | -1.15 (0.54) | -1.83 (0.58) | -2.13 (0.49)
  Visit 20 (Day 22) | -0.54 (0.29) | -1.54 (0.62) | -0.81 (0.44) | -1.27 (0.42) | -1.75 (0.53) | -2.19 (0.38)
  Visit 23 (Day 25) | -0.75 (0.42) | -1.81 (0.60) | -1.17 (0.55) | -1.46 (0.57) | -2.00 (0.42) | -2.21 (0.36)

5. Secondary Outcome: Change in Infiltration Compared to Baseline
Description: The severity of the symptoms was rated on screening and on study Days 1 (baseline), 4, 8, 11, 15, 18, 22, 25 and 29 (end of treatment) according to the 0-3 with half-point TCS grading scale.
  The (sub)investigator made the following clinical assessments by use of the scale below:
  Score; Intensity; Description
  Infiltration:
  0; No evidence 0.5; Doubtful or very mild 1.0; Mild Slight definite infiltration 1.5; Mild to moderate 2.0; Moderate; Moderate infiltration 2.5; Moderate to severe 3.0; Severe; Very marked infiltration
Time Frame: At Day 4, Day 8, Day 11, Day 15, Day 18, Day 22, and Day 25
Population: The 24 participants that were randomized received all products distributed on six different test sites on the body.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  Visit 5 (Day 4) | -0.06 (0.27) | -0.10 (0.29) | -0.04 (0.20) | 0.00 (0.21) | -0.27 (0.25) | -0.29 (0.33)
  Visit 8 (Day 8) | -0.06 (0.31) | -0.38 (0.34) | -0.13 (0.34) | -0.29 (0.51) | -0.73 (0.47) | -0.79 (0.44)
  Visit 11 (Day 11) | -0.13 (0.37) | -0.77 (0.51) | -0.31 (0.38) | -0.46 (0.39) | -1.06 (0.50) | -1.29 (0.62)
  Visit 14 (Day 15) | -0.25 (0.33) | -0.98 (0.60) | -0.42 (0.43) | -0.69 (0.38) | -1.35 (0.65) | -1.79 (0.59)
  Visit 17 (Day 18) | -0.33 (0.35) | -1.10 (0.61) | -0.58 (0.46) | -0.75 (0.39) | -1.50 (0.63) | -1.94 (0.61)
  Visit 20 (Day 22) | -0.31 (0.29) | -1.25 (0.66) | -0.56 (0.47) | -0.90 (0.33) | -1.67 (0.62) | -1.98 (0.52)
  Visit 23 (Day 25) | -0.38 (0.34) | -1.35 (0.73) | -0.73 (0.47) | -1.06 (0.40) | -1.67 (0.60) | -2.02 (0.54)

6. Secondary Outcome: Change in Total Clinical Score (TCS) of the Clinical Symptoms Compared to Baseline
Description: as for outcome 1
Time Frame: At Day 4, Day 8, Day 11, Day 15, Day 18, Day 22, and Day 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale
  Visit 5 (Day 4) | -0.27 (0.66) | -0.63 (0.80) | -0.19 (0.53) | -0.29 (0.66) | -1.00 (0.88) | -1.19 (0.86)
  Visit 8 (Day 8) | -0.42 (0.78) | -1.92 (1.18) | -0.88 (0.97) | -1.21 (1.07) | -2.81 (1.26) | -2.85 (1.17)
  Visit 11 (Day 11) | -0.75 (0.75) | -2.85 (1.26) | -1.40 (0.90) | -1.60 (1.11) | -3.71 (1.28) | -4.40 (1.42)
  Visit 14 (Day 15) | -1.17 (0.89) | -3.54 (1.66) | -1.75 (1.12) | -2.46 (1.00) | -4.48 (1.56) | -5.23 (1.41)
  Visit 17 (Day 18) | -1.42 (0.95) | -4.00 (1.72) | -2.23 (1.11) | -2.88 (0.99) | -5.04 (1.46) | -5.69 (1.30)
  Visit 20 (Day 22) | -1.31 (0.83) | -4.27 (1.92) | -2.21 (1.20) | -3.21 (0.98) | -5.17 (1.64) | -6.02 (1.08)
  Visit 23 (Day 25) | -1.54 (0.97) | -4.71 (1.99) | -2.75 (1.32) | -3.60 (1.25) | -5.50 (1.47) | -6.17 (0.87)

7. Secondary Outcome: Ultrasonography: Change in Lesions Thickness From Baseline Measured by Ultrasound
Description: The lesion thickness was measured by ultrasound at baseline, Day 8, Day 15, Day 22 and end of treatment.
Time Frame: At Day 8, Day 15, Day 22 and end of treatment
Population: The 24 participants that were randomized received all products distributed on six different test sites on the body.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- LEO 29102 Cream Vehicle: LEO 29102 cream vehicle without any active substance applied topically twice daily for 4 weeks.
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
mm
  Visit 8 (Day 8) | 0.05 (0.22) | -0.14 (0.32) | 0.03 (0.24) | 0.00 (0.24) | -0.30 (0.27) | -0.39 (0.30)
  Visit 14 (Day 15) | -0.05 (0.23) | -0.45 (0.39) | -0.16 (0.31) | -0.25 (0.36) | -0.51 (0.32) | -0.68 (0.46)
  Visit 20 (Day 22) | -0.07 (0.27) | -0.54 (0.37) | -0.15 (0.19) | -0.24 (0.32) | -0.57 (0.34) | -0.68 (0.39)
  Visit 26 (Day 29) | -0.13 (0.30) | -0.63 (0.39) | -0.30 (0.31) | -0.38 (0.30) | -0.68 (0.34) | -0.78 (0.43)

8. Secondary Outcome: Biomarkers by Immunochemistry
Description: 3 skin biopsies (punch biopsies of 3 mm) per participant were taken on Day 29 after the clinical scoring and ultrasound measurement.
  Cells counted per mm^2 were cells that were positive for the indicated biomarker.
Time Frame: At end of treatment
Population: Since biopsies were only taken from three out of six sites, not all treatment-block combinations were available.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
cells/mm^2
  Macrophages: CD163: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  Macrophages: CD163 | 313.9 (97.28) | 197.4 (69.51) | 291.2 (100.8) | 383.5 (488.6) | 178.2 (27.96) | 172.9 (40.61)
  Dendritic cells CD1a: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  Dendritic cells CD1a | 233.8 (113.9) | 42.14 (27.81) | 229.3 (134.2) | 244.0 (118.9) | 34.31 (20.00) | 56.34 (33.81)
  T-cell biomarker CD3: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  T-cell biomarker CD3 | 593.8 (243.9) | 124.5 (105.9) | 464.2 (275.9) | 492.7 (280.4) | 126.1 (95.57) | 143.9 (161.5)
  Angiogenesis: CD31: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  Angiogenesis: CD31 | 430.7 (165.7) | 216.3 (100.1) | 331.1 (120.9) | 348.8 (158.1) | 184.2 (38.84) | 186.6 (51.62)
  T-cell biomarker: CD4: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  T-cell biomarker: CD4 | 284.3 (123.9) | 59.17 (41.78) | 246.4 (148.0) | 239.0 (147.3) | 55.56 (44.03) | 66.95 (55.07)
  T-cell biomarker: CD45RO: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  T-cell biomarker: CD45RO | 752.0 (183.1) | 101.6 (78.14) | 630.1 (318.8) | 643.6 (370.4) | 121.6 (50.39) | 218.2 (258.7)
  Macrophages: CD68: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  Macrophages: CD68 | 370.8 (58.56) | 120.3 (61.57) | 323.1 (114.2) | 303.8 (117.8) | 142.1 (58.47) | 156.8 (44.82)
  T-cell biomarker: CD8: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  T-cell biomarker: CD8 | 280.5 (156.0) | 60.05 (61.95) | 220.7 (123.9) | 253.2 (171.9) | 66.35 (53.30) | 65.05 (72.00)

9. Secondary Outcome: Biomarkers by Immunochemistry: Epidermal Differentiation
Description: 3 skin biopsies (punch biopsies of 3 mm) per participant were taken on Day 29 after the clinical scoring and ultrasound measurement.
Time Frame: At end of treatment
Population: Since biopsies were only taken from three out of six sites, not all treatment-block combinations were available.
Measure: Mean (Standard Deviation); unit: %, positive area/total area
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
%, positive area/total area
  Epidermal differentiation: CK10: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  Epidermal differentiation: CK10 | 0.76 (0.14) | 0.89 (0.15) | 0.77 (0.14) | 0.75 (0.11) | 0.93 (0.08) | 0.89 (0.25)
  Epidermal differentiation: CK16: number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
  Epidermal differentiation: CK16 | 0.11 (0.14) | 0.00 (0.00) | 0.08 (0.11) | 0.02 (0.04) | 0.01 (0.01) | 0.00 (0.01)

10. Secondary Outcome: Biomarkers by Immunochemistry: Epidermal Proliferation
Description: 3 skin biopsies (punch biopsies of 3 mm) per participant were taken on Day 29 after the clinical scoring and ultrasound measurement.
  By measurement of the cell-cycle marker, Ki-67 protein, an evaluation of the degree of skin cell proliferation and thereby epidermal proliferation could be obtained. Cells counted per mm^2 were cells that were positive for the indicated biomarker.
Time Frame: At end of treatment
Population: Since biopsies were only taken from three out of six sites, not all treatment-block combinations were available.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
cells/mm^2 | 554.1 (391.9) | 19.45 (28.69) | 443.3 (298.6) | 354.3 (198.2) | 20.50 (29.11) | 93.49 (134.9)

11. Secondary Outcome: Pathology and Histology by Treatment
Description: Skin biopsies were taken on Day 29. The evaluation of immunohistochemical sections were performed on cross sections of the skin tissue. The same pathologist did all evaluations, and samples were masked to ensure a blind fashion study. The extent of the following parameters were measured in scored semi-quantitatively (semi) on blinded haematoxylin and eosin (HE) sections. Semi-quantitative scoring was categorized as No (0), mild (1), moderate (2), marked (3) or severe (4). In evaluating the morphology of epidermis (Stratum corneum and Stratum granulosum) the tissue was classified by the characteristics seen below:
  * Morphology of epidermis
    * Stratum corneum (semi (extent of))
    * Stratum granulosum (semi (extent of))
    * Parakeratosis (semi (extent of))
  * Infiltration of inflammatory cells (semi (extent of))
Time Frame: At end of treatment
Population: Since biopsies were only taken from three out of six sites, not all treatment-block combinations were available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale
  Infiltration of inflammatory cells: number analyzed (Participants) | 12 | 6 | 23 | 17 | 6 | 6
  Infiltration of inflammatory cells | 1.50 (0.80) | 0.17 (0.41) | 1.52 (0.79) | 1.53 (0.94) | 0.50 (0.55) | 0.67 (1.03)
  Parakeratosis: number analyzed (Participants) | 12 | 6 | 23 | 17 | 6 | 6
  Parakeratosis | 1.67 (1.15) | 0.00 (0.00) | 1.39 (1.34) | 1.35 (1.11) | 0.00 (0.00) | 0.17 (0.41)
  Stratum Corneum: number analyzed (Participants) | 12 | 6 | 23 | 17 | 6 | 6
  Stratum Corneum | 1.83 (0.83) | 0.33 (0.52) | 1.52 (0.90) | 1.41 (0.94) | 0.50 (0.55) | 0.33 (0.82)
  Stratum Granulosum: number analyzed (Participants) | 12 | 6 | 23 | 17 | 6 | 6
  Stratum Granulosum | 1.42 (1.24) | 0.17 (0.41) | 1.04 (1.26) | 1.00 (1.17) | 0.00 (0.00) | 0.17 (0.41)

12. Secondary Outcome: Pathology and Histology by Treatment: Epidermal Thickness
Description: Skin biopsies were taken on Day 29. The evaluation of immunohistochemical sections were performed on cross sections of the skin tissue. The same pathologist did all evaluations, and samples were masked to ensure a blind fashion study. In evaluating the morphology of epidermis (Stratum corneum and Stratum granulosum), the tissue was classified by the characteristic epidermal thickness. This was measured in the absolute number of µm measured on blinded haematoxylin and eosin (HE) sections..
Time Frame: At end of treatment
Population: Since biopsies were only taken from three out of six sites, not all treatment-block combinations were available.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 12 | 6 | 24 | 18 | 6 | 6
µm | 254.6 (58.68) | 73.81 (20.61) | 187.5 (79.65) | 176.4 (49.05) | 68.48 (18.16) | 66.90 (44.53)

13. Secondary Outcome: Pathology and Histology by Treatment: Frequency of Neutrophil Abscesses
Description: Skin biopsies were taken on Day 29. The evaluation of immunohistochemical sections were performed on cross sections of the skin tissue. The same pathologist did all evaluations, and samples were masked to ensure a blind fashion study.
  In evaluating the morphology of epidermis (Stratum corneum and Stratum granulosum), the tissue was classified by the characteristic of frequency of neutrophil microabscesses (Monroe´s abscess). This was measured in absolute number of cells that were positive for the marker on blinded haematoxylin and eosin (HE) sections.
Time Frame: At end of treatment
Population: Since biopsies were only taken from three out of six sites, not all treatment-block combinations were available.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | LEO 29102 Cream Vehicle | Betamethasone Dipropionate Cream | LEO 29102 Cream | LEO 29102 Plus Calcipotriol Cream | LEO 29102 Plus Betamethasone Dipropionate | Daivobet® Ointment
Number analyzed (Participants) | 11 | 6 | 23 | 17 | 6 | 6
cells/mm^2 | 0.14 (0.26) | 0.00 (0.00) | 0.15 (0.35) | 0.17 (0.30) | 0.00 (0.00) | 0.05 (0.13)

ADVERSE EVENTS:
Time Frame: From baseline to end of Follow-up (Day 43±2)
Arm/Group | All Randomized Participants
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Randomized Participants (N=24)
Diarrhoea (Gastrointestinal disorders) | 3
Diverticulitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Hordeolum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Postoperative infection (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO retains the right to publish the results of this clinical trial.